CLINICAL TRIAL: NCT01325272
Title: Interrelations Between Spontaneous Otoacoustic Emissions and Transient Evoked Emissions: Indication of Cochlear Damage in Newborn.
Brief Title: Interrelations Between Spontaneous Otoacoustic Emissions and Transient Evoked Emissions
Status: Completed | Type: Observational
Sponsor: UPECLIN HC FM Botucatu Unesp (Other)
Responsible Party: Daniela Polo Camargo da Silva, Faculdade de Medicina de Botucatu
Other Study IDs: upeclin/HC/FMB-Unesp-53
Record Dates: First submitted 2011-03-28; First posted 2011-03-29 (Estimated); Last update posted 2011-06-01 (Estimated); Status verified 2011-05

CONDITIONS: Cochlear Function
Keywords: otoacoustic emissions in newborns

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- preterm newborn
- term newborn

SUMMARY:
To verify the occurrence of Spontaneous Otoacoustic Emissions (SOAE) in neonates at term and preterm infants who had transient otoacoustic emissions and verify if the presence of response is related to gestational age, gender or risk factors for hearing loss.

ELIGIBILITY:
Inclusion Criteria:

* born in this institution
* have presence of transient otoacoustic emission

Exclusion Criteria:

-

Ages: 4 Days to 5 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children born in this institution
Sampling Method: Probability Sample
Dates: Start 2009-03; Study Completion 2009-09

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Polo Camargo da Silva, Mestre, Principal Investigator — Faculdade de Medicina de Botucatu
Locations (1):
- Faculdade de Medicina de Botucatu, Botucatu, São Paulo, Brazil